CLINICAL TRIAL: NCT00896207
Title: Single-Dose Phase 0 Exploratory Pharmacokinetic Clinical Trial Comparing Five Oral Formulations of SR13668, an Orally Active AKT Pathway Inhibitor
Brief Title: Studying Different Formulations of SR13668 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01106; NCI-2009-01106 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MAYO-MAY07-9-01; CDR0000638390; MAY-07-9-01; MAYO-MAY07-9-01 (Other: Mayo Clinic); MAY07-9-01 (Other: DCP); P30CA015083 (NIH)
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2011-10

CONDITIONS: Healthy, no Evidence of Disease

ARMS (6):
- Arm I (Experimental): Participants complete an overnight fast of ≥ 10 hours, eat a high-fat (approximately 50% of total caloric content of the meal) and high-calorie (approximately 800-1,000 calories) meal, and then receive a single dose of oral SR13668 in a PEG400/Labrasol® liquid formulation with 8 ounces of water. Participants may not eat for ≥ 4 hours after study drug administration.
  Interventions: Drug: Akt inhibitor SR13668
- Arm II (Experimental): Participants complete an overnight fast of ≥ 10 hours and then receive a single dose of oral SR13668 in a PEG400/Labrasol® liquid formulation with 8 ounces of water. Participants may not eat for ≥ 4 hours after study drug administration.
  Interventions: Drug: Akt inhibitor SR13668
- Arm III (Experimental): Participants receive a single dose of oral Akt inhibitor SR13668 in a Solutol® self-emulsifying solid dispersion capsule formulation.
  Interventions: Drug: Akt inhibitor SR13668
- Arm IV (Experimental): Participants receive a single dose of oral Akt inhibitor SR13668 in a Solutol®/vitamin E TGPS self-emulsifying solid dispersion capsule formulation.
  Interventions: Drug: Akt inhibitor SR13668
- Arm V (Experimental): Participants receive a single dose of oral Akt inhibitor SR13668 in a vitamin E TGPS self-emulsifying solid dispersion capsule formulation.
  Interventions: Drug: Akt inhibitor SR13668
- Arm VI (Experimental): Participants receive a single dose of oral Akt inhibitor SR13668 in a Myrj 53 self-emulsifying solid dispersion capsule formulation.
  Interventions: Drug: Akt inhibitor SR13668

INTERVENTIONS:
Drug: Akt inhibitor SR13668 — Given orally as a single dose
  Other Names: SRI13668

SUMMARY:
This randomized early phase I trial is studying different formulations of SR13668 in healthy volunteers. Giving SR13668 may help doctors learn more about how SR13668 is used by the body. It is not yet known which formulation of SR13668 is most effectively used by the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine which oral formulation of Akt inhibitor SR13668 provides the best bioavailability in normal, healthy volunteers.

SECONDARY OBJECTIVES:

I. Determine the oral pharmacokinetics of a single, low dose of Akt inhibitor SR13668 in healthy volunteers.

II. Characterize the metabolism of Akt inhibitor SR13668 in healthy volunteers. III. Collect preliminary safety data for Akt inhibitor SR13668 in healthy volunteers.

OUTLINE:

STAGE 1 (for the first 6 participants enrolled in the study [closed to accrual as of August, 2009]): Participants are randomized to 1 of 2 arms.

ARM I: Participants complete an overnight fast of ≥ 10 hours, eat a high-fat (approximately 50% of total caloric content of the meal) and high-calorie (approximately 800-1,000 calories), and then receive a single dose of oral SR13668 in a PEG400/Labrasol® liquid formulation with 8 ounces of water. Participants may not eat for ≥ 4 hours after study drug administration.

ARM II: Participants complete an overnight fast of ≥ 10 hours and then receive a single dose of oral SR13668 in a PEG400/Labrasol® liquid formulation with 8 ounces of water. Participants may not eat for ≥ 4 hours after study drug administration.

STAGE 2 (for the next 12 participants enrolled in the study): The preferred dietary condition (Arm I) identified in stage 1 is used. Participants are randomized to 1 of 4 arms.

ARM III: Participants receive a single dose of oral Akt inhibitor SR13668 in a Solutol® self-emulsifying solid dispersion capsule formulation.

ARM IV: Participants receive a single dose of oral Akt inhibitor SR13668 in a Solutol®/vitamin E TGPS self-emulsifying solid dispersion capsule formulation.

ARM V: Participants receive a single dose of oral Akt inhibitor SR13668 in a vitamin E TGPS self-emulsifying solid dispersion capsule formulation.

ARM VI: Participants receive a single dose of oral Akt inhibitor SR13668 in a Myrj 53 self-emulsifying solid dispersion capsule formulation.

Blood and urine samples are collected at baseline and periodically during the 24 hours after study drug administration for pharmacokinetic analysis by high performance liquid chromatography assay.

After completion of study treatment, participants are followed by telephone at 7-10 days and at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* ECOG performance status 0
* Leukocyte count ≥ 3,000/mm^3
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin normal
* Alkaline phosphatase ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 1.5 times ULN
* Direct bilirubin ≤ 1.5 times ULN
* Sodium ≤ 1.5 times ULN
* Potassium ≤ 1.5 times ULN
* Creatinine ≤ 1.5 times ULN OR calculated creatinine clearance ≥ 30 mL/min
* Fasting blood glucose normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile participants must use effective barrier contraception
* Able and willing to fast overnight prior to study drug administration AND consume a high-fat meal on the day of study drug administration
* Willing to provide required blood and urine samples AND stay all day and overnight in the Clinical Research Unit
* Willing to abstain from alcoholic beverages and caffeine for ≥ 24 hours prior to study drug administration and until all blood and urine samples have been collected
* No cancer within the past 3 years except for nonmelanoma skin cancer, localized prostate cancer, superficial bladder cancer, or carcinoma in situ of the cervix
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Severe chronic obstructive pulmonary disease requiring supplemental oxygen
  * Hypertension that is difficult to control
  * Psychiatric illness or social situation that would limit compliance with study requirements
* No diabetes mellitus
* No other condition that may, in the investigator's opinion, interfere with ingestion or absorption of oral medications (e.g., inflammatory bowel disease)
* No history of allergic-type reactions, including asthma and urticaria, or other intolerance to chemical compounds similar to the active study agent, indole-3-carbinol, or cruciferous vegetables (e.g., cabbage, cauliflower, broccoli, kale, and Brussels sprouts)
* More than 6 months since prior investigational agents
* More than 3 months since prior oral contraceptives (including Plan B method of contraception)

  * No concurrent hormonal contraception
* More than 14 days since prior and no concurrent anticoagulant or antiplatelet medications
* More than 7 days since prior and no concurrent daily medications or nutritional supplements
* No prior gastrectomy that may, in the investigator's opinion, interfere with ingestion or absorption of oral medications
* No other concurrent medications

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Food effect on the bioavailability of SR13668 after oral administration | Up to 30 days after completion of study treatment
  The first stage will be used to compare fed vs. fasted diet effect on the pharmacokinetics parameters under formulation 1.
Formulation effect on the bioavailability of SR13668 after oral administration | Up to 30 days after completion of study treatment
  The second stage will be used to determine the formulation effects on the pharmacokinetics parameters, all under either fed or fasted diet as determined by the first stage.

SECONDARY OUTCOMES:
Solubility and stability of Akt inhibitor SR13668 in oral formulations selected for exploratory pharmacokinetics studies | Up to 30 days after completion of study treatment
Oral pharmacokinetics of a single low dose of Akt inhibitor SR13668 | Up to 30 days after completion of study treatment
Metabolism of Akt inhibitor SR13668 | Up to 30 days after completion of study treatment
Preliminary safety data for Akt inhibitor SR13668, graded according to NCI CTCAE version 3.0 | Up to 30 days after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paul Limburg, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States